CLINICAL TRIAL: NCT04598399
Title: Comparison of the Effectiveness of Two Psycho-physical Interventions: Mindfulness Based Relapse Prevention (MBRP) and Unguided Meditative Relaxation in Patients With Alcohol Use Disorder
Acronym: MBRP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PHRCN/2018/AL-01
Record Dates: First submitted 2020-10-16; First posted 2020-10-22 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Alcohol Use Disorder (AUD)
MeSH Terms: conditions — Alcoholism | interventions — Meditation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: In order to limit measurement and attrition biases, the patient will be kept unaware of the hypotheses concerning the details of the evaluated programs (MBRP or control) and the program expected to be superior
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MBRP program: (Experimental)
  Interventions: Behavioral: Mindfulness Based Relapse Prevention
- Standard care (Active Comparator)
  Interventions: Behavioral: Relaxation/ meditation

INTERVENTIONS:
Behavioral: Mindfulness Based Relapse Prevention — 7 x 60-120 minute sessions with different themes: Automatic pilot/triggers/relapse/high-risk situations/ mindfulness in daily life. There will be a welcoming time, with a focus on at-home practice and difficulties, a theoretical presentation of new concepts, practical meditation exercises and a debriefing.
  Arms: MBRP program:
Behavioral: Relaxation/ meditation — 7 x 60-120 minute sessions each with a different sound from nature with unguided, closed relaxation group with a maximum of 12 participants
  Arms: Standard care

SUMMARY:
Alcohol use disorder (AUD) is the second highest preventable cause of death in France. Only 3% of patients are prescribed approved drugs for reducing alcohol consumption or maintenance of abstinence. Increasing evidence supports the efficacy of psychotherapies such as cognitive and behavioral therapies (CBT) in AUD. However, some patients are resistant to CBT and the positive effects of CBT could wane over time, resulting in mid- and long-term relapses. Mindfulness practice is increasingly widespread in the United States and its efficacy in various fields appears very promising. The study investigators hypothesize that the Mindfulness Based Relapse Prevention (MBRP) program will be more efficient than a relaxation/meditation without guidance control program in AUD.

ELIGIBILITY:
Inclusion Criteria:

* Having a moderate to severe alcohol use disorder according to DSM 5 criteria.
* The last drink must have been consumed at most in the last 60 days before the pre-inclusion visit. The patient must have had at least 1 HDD during the last drinking period

Exclusion Criteria:

* Severe depression (Beck Depression Inventory> 30)
* Schizophrenic disorder,
* Current maniac or hypomaniac episode,
* Patient with dementia or severe cognitive impairment that would prevent him/her from following the course of a session, as judged by the clinician.
* Insufficient French understanding to complete the questionnaires
* Pregnant or breastfeeding woman
* Absence of social security regimen
* Other mindfulness-based structured therapies
* Refusal to sign the written consent. • The patient is under safeguard of justice or state guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in number of heavy drinking days (HDD) over previous 4 weeks, between the last drinking period at inclusion and 6 months. | 6 months
  Alcohol Time Line Follow Back (TLFB) where a HDD = consummation of 4+ (for women) or 5+ (for men) drinks per day.

SECONDARY OUTCOMES:
Change in number of heavy drinking days (HDD) during the last 4 weeks, between the last drinking period at inclusion and 3 months between groups | 3 months
  Alcohol Time Line Follow Back (TLFB) where a HDD = consummation of 4+ (for women) or 5+ (for men) drinks per day.
Change in number of heavy drinking days (HDD) during the last 4 weeks, between the last drinking period at inclusion and 12 months between groups | 12 months
  Alcohol Time Line Follow Back (TLFB) where a HDD = consummation of 4+ (for women) or 5+ (for men) drinks per day.
Change in 4-week total alcohol consumption since baseline | 3 months
  number of drinks (1 glass = 1 unit according to grams alcohol)
Change in 4-week total alcohol consumption since baseline | 12 months
  number of drinks (1 glass = 1 unit according to grams alcohol)
Change in frequency of craving since baseline | 3 months
  version F of craving experience questionnaire (CEQ-F)
Change in frequency of craving since baseline | 6 months
  version F of craving experience questionnaire (CEQ-F)
Change in frequency of craving since baseline | 12 months
  version F of craving experience questionnaire (CEQ-F)
Change in strength of craving since baseline | 3 months
  version S of craving experience questionnaire (CEQ-S)
Change in strength of craving since baseline | 6 months
  version S of craving experience questionnaire (CEQ-S)
Change in strength of craving since baseline | 12 months
  version S of craving experience questionnaire (CEQ-S)
Anxiety at baseline | Baseline
  Beck Anxiety Inventory depression (BAI): 21-item self-assessment scale assessing anxiety
Change in anxiety since baseline | 3 months
  Beck Anxiety Inventory depression (BAI): 21-item self-assessment scale assessing anxiety
Change in anxiety since baseline | 6 months
  Beck Anxiety Inventory depression (BAI): 21-item self-assessment scale assessing anxiety
Change in anxiety since baseline | 12 months
  Beck Anxiety Inventory depression (BAI): 21-item self-assessment scale assessing anxiety
Depression at baseline | Baseline
  Beck Depression Inventory (BDI): 21 items assessing the presence and severity of depressive symptoms
Change in depression since baseline | 3 months
  Beck Depression Inventory (BDI): 21 items assessing the presence and severity of depressive symptoms
Change in depression since baseline | 6 months
  Beck Depression Inventory (BDI): 21 items assessing the presence and severity of depressive symptoms
Change in depression since baseline | 12 months
  Beck Depression Inventory (BDI): 21 items assessing the presence and severity of depressive symptoms
Change in quality of life since baseline | 3 months
  Alcohol Quality of Life Scale (AQoLS): 34-item patient-reported questionnaire
Change in quality of life since baseline | 6 months
  Alcohol Quality of Life Scale (AQoLS): 34-item patient-reported questionnaire
Change in quality of life since baseline | 12 months
  Alcohol Quality of Life Scale (AQoLS): 34-item patient-reported questionnaire
Emotion regulation at baseline | Baseline
  Emotion Regulation Questionnaire (ERQ): 10-item scale designed to assessing Cognitive Reappraisal and Expressive Suppression on a 7-point Likert-type scale ranging from 1 (strongly disagree) to 7 (strongly agree).
Change in emotion regulation since baseline | 3 months
  Emotion Regulation Questionnaire (ERQ): 10-item scale designed to assessing Cognitive Reappraisal and Expressive Suppression on a 7-point Likert-type scale ranging from 1 (strongly disagree) to 7 (strongly agree).
Change in emotion regulation since baseline | 6 months
  Emotion Regulation Questionnaire (ERQ): 10-item scale designed to assessing Cognitive Reappraisal and Expressive Suppression on a 7-point Likert-type scale ranging from 1 (strongly disagree) to 7 (strongly agree).
Change in emotion regulation since baseline | 12 months
  Emotion Regulation Questionnaire (ERQ): 10-item scale designed to assessing Cognitive Reappraisal and Expressive Suppression on a 7-point Likert-type scale ranging from 1 (strongly disagree) to 7 (strongly agree).
Difficulties regulating emotion at baseline | Baseline
  Difficulties in Emotion Regulation scale (DERS -Impulse): items 3, 14, 19, 24R, 27, 32 from DERS
Changes in difficulties regulating emotion since baseline | 3 months
  Difficulties in Emotion Regulation scale (DERS -Impulse): items 3, 14, 19, 24R, 27, 32 from DERS
Changes in difficulties regulating emotion since baseline | 6 months
  Difficulties in Emotion Regulation scale (DERS -Impulse): items 3, 14, 19, 24R, 27, 32 from DERS
Changes in difficulties regulating emotion since baseline | 12 months
  Difficulties in Emotion Regulation scale (DERS -Impulse): items 3, 14, 19, 24R, 27, 32 from DERS
Changes in impulsivity since baseline | 3 months
  Impulsive behavior scale (UPPS-P): 20-item self-assessment scale
Impulsivity at baseline | Baseline
  Impulsive behavior scale (UPPS-P): 20-item self-assessment scale
Changes in impulsivity since baseline | 6 months
  Impulsive behavior scale (UPPS-P): 20-item self-assessment scale
Changes in impulsivity since baseline | 12 months
  Impulsive behavior scale (UPPS-P): 20-item self-assessment scale
Changes in coping mechanism | 3 months
  brief COPE questionnaire: 14 scales including 2 items (28 items in total)
Coping mechanism at baseline | Baseline
  brief COPE questionnaire: 14 scales including 2 items (28 items in total)
Changes in coping mechanism | 6 months
  brief COPE questionnaire: 14 scales including 2 items (28 items in total)
Changes in coping mechanism | 12 months
  brief COPE questionnaire: 14 scales including 2 items (28 items in total)
Cognitive impairment | Baseline
  Montreal Cognitive Assessment (MoCA)
Initial mindfulness | Baseline
  Five Facets Mindfulness Questionnaire (FFMQ): 39-item self-assessment tool measuring 5 factors of mindfulness
Number of meditation sessions per week over the last 4 weeks | Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Amandine Luquiens, Principal Investigator — CHU Nimes
Locations (7):
- France (7):
  - Ssra Les Eumenides, Angers
  - Hôpital Corentin-Celton, Issy-les-Moulineaux
  - CHU de Nantes, Nantes
  - CHU de Nimes, Nîmes
  - Hopital Fernand Widal, Paris
  - Hopital Des 4 Villes, Sèvres
  - Hopital Paul Brousse, Villejuif

IPD SHARING:
Plan to Share IPD: No